CLINICAL TRIAL: NCT05338411
Title: Effect of Exogenous Growth Hormone on Ocular Findings of Children With Precocious and Early Puberty: a Prospective Cohort Study
Brief Title: Effect of Exogenous Growth Hormone on Ocular Findings
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohsen Pourazizi, Dr. Mohsen Pourazizi, Isfahan University of Medical Sciences
Other Study IDs: IR.ARI.MUI.REC.1400.121
Record Dates: First submitted 2022-04-10; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Precocious Puberty; Early Puberty; Refraction Error
Keywords: Precocious Puberty; Early Puberty; human growth hormone; Refraction Error; Axial Length
MeSH Terms: conditions — Puberty, Precocious; Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Early or precocious puberty who receive GH: Children with early or precocious puberty who receive exogenous growth hormone
- Early or precocious puberty who does not receive GH: Children with early or precocious puberty who does not receive exogenous growth hormone
- Healthy: Healthy children without any past medical history

SUMMARY:
Body size and eye function play an essential role in adapting to the environment and human survival. Growth hormone is commonly recognized by its effect on the height of individuals; Although from an evolutionary perspective, the effects of growth hormone on eye development are more important. Although the effect of growth hormone on eye development has not been accurately determined, the results of a number of studies suggest the effect of growth hormone on eye development.

Despite the large number of studies that have investigated the effects of growth hormone on height growth, there are few studies that have investigated the effects of growth hormone on the eye.

To the best of our knowledge, no study has been conducted to investigate the effect of growth hormone on ocular findings of patients with early or precocious puberty. Therefore, we intend to investigate the effect of growth hormone on ocular findings of patients with early or precocious puberty.

DETAILED DESCRIPTION:
Investigators will achieve the following data from the participants:

1. Demographics
2. Past medical history

3. Bone and calendar age

4- Stage of puberty

5- Ocular examination

6. Ocular biometry

ELIGIBILITY:
Inclusion Criteria:

Sample group (with early or precocious puberty):

1. Children with precocious puberty based on Tanner classification
2. Girls 4 to 10 years old
3. Boys aged 4 to 11
4. No known eye problems including: history of eye trauma, eye surgery 5- lack of family history of glaucoma or increased intraocular pressure

6. Lack of previous history of receiving growth hormone 7. Lack of systemic disease or known syndromes 8. Consent to participate in the study

Exclusion Criteria:

1. Incidence of growth hormone adverse reactions leading to discontinuation of treatment
2. Changing the patient's treatment plan during the study
3. Ocular complications requiring treatment during the study
4. Unwillingness of the patient to continue participating in the study

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study groups are children with early or precocious puberty referred to endocrine clinic of Imam Hossein Hospital in Isfahan, Iran. The control group will be selected from the children who visit at the health centers for routine examinations.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-03-20 (Actual); Primary Completion 2023-10-22 (Estimated); Study Completion 2023-10-22 (Estimated)

PRIMARY OUTCOMES:
Refraction Error | 6 months
  Comparison of the refraction error between the study groups
Axial Length | 6 months
  Comparison of the axial length between the study groups

SECONDARY OUTCOMES:
Papillitis | 6 months
  Comparison of the frequency of papillitis between the study groups
Central Corneal Thickness | 6 months
  Comparison of the mean central corneal thickness between the study groups

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - Isfahan University of Medical Sciences, Isfahan
  - Isfahan Eye Research Center, Isfahan